CLINICAL TRIAL: NCT06642987
Title: An Open-label, Randomized, Fasting, Single-dose, 2x2, Crossover Study in Healthy Subjects to Evaluate the Bioequivalence of Vonopzan Tablets 20mg(Vonoprazan Fumarate) of Hanlim and Vocinti Tablet 20mg(Vonoprazan Fumarate) of Takeda.
Brief Title: Study to Evaluate the Bioequivalence of Vonopzan Tablet 20mg(Vonoprazan Fumarate) and Vocinti Tablet 20mg in Healthy Adult Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DDS23-018BE
Record Dates: First submitted 2024-10-14; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Gastric Ulcer
MeSH Terms: conditions — Stomach Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vonoprazan Test 20mg (Experimental): On the day of the visit, take 1 tablet of the experimental drug orally with 150 mL of water around 8 am.
  Interventions: Drug: Vonoprazan Test 20mg
- Vonoprazan Reference 20mg (Active Comparator): On the day of the visit, take 1 tablet of the comparator drug orally with 150 mL of water around 8 am.
  Interventions: Drug: Vonoprazan Reference 20mg

INTERVENTIONS:
Drug: Vonoprazan Test 20mg — 1 tablets orally once a day
  Other Names: vonoprazan fumarate
  Arms: Vonoprazan Test 20mg
Drug: Vonoprazan Reference 20mg — 1 tablets orally once a day
  Other Names: Vonoprazna fumarate
  Arms: Vonoprazan Reference 20mg

SUMMARY:
This clinical trial is an open-label, randomized, fasting, single-dose, two-sequence, two-period, crossover study in healthy subjects to evaluate the bioequivalence of "Vonopzan Tablets 20 mg(Vonoprazan Fumarate)" of Hanlim Pharm.l Co., Ltd. and "Vocinti Tablet 20 mg (Vonoprazan Fumarate)" of Takeda Pharmaceuticals Korea Co., Ltd. in Healthy Adult Subjects.

DETAILED DESCRIPTION:
This study is to compare and evaluate the safety and pharmacokinetic characteristics of "Vonopzan Tablets 20 mg(Vonoprazan Fumarate)" of Hanlim Pharm. Co., Ltd. as the test drug and "Vocinti Tablet 20 mg (Vonoprazan Fumarate)" of Takeda Pharmaceuticals Korea Co., Ltd. as the reference drug in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 19 years or older at the time of screening
2. Individuals with no clinically significant congenital or chronic diseases and no pathological symptoms or findings based on medical examinations (such as EEG, ECG, chest and gastric endoscopy, or gastrointestinal radiology tests, if necessary)
3. Individuals deemed suitable for the study based on screening tests (e.g., hematology, blood chemistry, serology, and urinalysis) as determined by the principal investigator (or a designated sub-investigator)
4. Individuals with a Body Mass Index (BMI) between 18.0 and 30.0 (BMI calculation: weight (kg) / height (m)²)
5. Individuals with no history of gastrointestinal surgery that could affect drug absorption.
6. Individuals who, after receiving a detailed explanation of the clinical trial, fully understand the study, voluntarily decide to participate, and agree in writing to comply with the trial requirements during the study period.

Exclusion Criteria:

1. Individuals who have taken enzyme-inducing or inhibiting drugs such as barbiturates within 30 days before the start of the study (first dosing day) or medications that might interfere with the study within 10 days before the start of the study (first dosing day)
2. Individuals who have engaged in excessive alcohol consumption within one month before the start of the study (first dosing day)

   * For men, more than an average of 21 drinks per week
   * For women, more than an average of 14 drinks per week (One drink: 45 mL of distilled spirits or 360 mL of beer or 150 mL of wine)
3. Individuals who have taken any medication that may interfere with the trial within 10 days prior to the start of the trial (first dose).
4. Individuals who have participated in clinical trials (including bioequivalence studies) and received investigational drugs within six months before the start of the study (first dosing day)
5. Individuals who have donated whole blood within 8 weeks or donated blood components within 2 weeks before the start of the study (first dosing day)
6. Patients with the following conditions:

   * Hypersensitivity to the components of this drug
   * Currently taking medications containing atazanavir, nelfinavir, or rilpivirine.
7. Individuals with a history of mental illness
8. Women who may be pregnant, pregnant women, or brestfeeding women
9. Individuals who do not agree to use medically recognized dual contraception* methods, excluding hormonal contraceptives, to prevent pregnancy from the first administration of the investigational drug until one week after the last administration of the investigational drug.

   - Medically recognized dual contraception methods: Combining intrauterine devices (IUD, IUS), vasectomy, tubal ligation, and barrier methods of contraception (male condom, female condom, cervical cap, diaphragm, sponge, etc.), or using two or more barrier methods in combination with spermicides.
10. Individuals deemed unsuitable for this clinical trial for reasons other than the above inclusion/exclusion criteria by the principal investigator (or a designated sub-investigator)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 36 hours
  Concentration of vonoprazan in plasma
Area under the plasma concentration versus time curve (AUC) | 36 hours
  Concentration of vonoprazan in plasma

SECONDARY OUTCOMES:
AUCt/AUC∞ | 36 hours
  Concentration of vonoprazan in plasma
Half life | 36 hours
  Concentration of vonoprazan in plasma
Tmax | 36 hours
  Concentration of vonoprazan in plasma
AUC ∞ | 36 hours
  Concentration of vonoprazan in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Seok Gyeong Medical Foundation Central Hospital, Siheung-si, South Korea